CLINICAL TRIAL: NCT00962663
Title: A Randomized, Placebo-Controlled, 3-way Crossover Study to Investigate the Pharmacodynamic Effects of ICA-105665 Using the Intradermal Capsaicin and UV-B Models in Healthy Male Subjects
Brief Title: Effects of ICA-105665 Using the Intradermal Capsaicin and Ultraviolet B (UV-B) Models in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: ICA-105665-05; B5311006
Record Dates: First submitted 2009-08-19; First posted 2009-08-20 (Estimated); Last update posted 2012-09-28 (Estimated); Status verified 2012-09

CONDITIONS: Healthy
MeSH Terms: interventions — Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- ICA-105665 (Experimental): Three study drug treatments will be used: ICA-105665, ibuprofen, and placebo (for both ICA-105665 and Ibuprofen). The order of study drug treatment given to each subject during each specified treatment period is determined at randomization.
  Interventions: Drug: ICA-105665
- Ibuprofen (Active Comparator): Three study drug treatments will be used: ICA-105665, ibuprofen, and placebo (for both ICA-105665 and Ibuprofen). The order of study drug treatment given to each subject during each specified treatment period is determined at randomization.
  Interventions: Drug: Ibuprofen
- Placebo (Placebo Comparator): Three study drug treatments will be used: ICA-105665, ibuprofen, and placebo (for both ICA-105665 and Ibuprofen). The order of study drug treatment given to each subject during each specified treatment period is determined at randomization.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ICA-105665 — Subjects randomized to receive ICA -105665 will receive 200 mg BID
  Arms: ICA-105665
Drug: Ibuprofen — Subjects randomized to receive Ibuprofen will receive placebo to ICA-105665 at all scheduled dosing times on Days 1 to 4 and a single dose of 800 mg Ibuprofen on the morning of Day 4.
  Other Names: Cuprofen
  Arms: Ibuprofen
Drug: Placebo — Subjects randomized to receive placebo will receive placebo to ICA
  -105665 at all scheduled dosing times on Days 1 to 4 and placebo to Ibuprofen on the morning of Day 4.
  Other Names: orange Syrup BP
  Arms: Placebo

SUMMARY:
The purpose of this study is; to determine the pharmacodynamic (PD) effects of ICA-105665 using the intradermal (ID) capsaicin model in healthy male subjects, and to investigate the effect of ICA-105665 on inflammatory hyperalgesia using the ultraviolet B (UV-B) model in healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males aged 18 to 55 years (inclusive).
* Body mass index (BMI) of 18 to 30 kg/m2.
* Non-smokers and smokers of up to 5 cigarettes or equivalent per day.
* Must be able to abstain from smoking during residential periods.
* Demonstration of positive hyperalgesia as defined by an area of hyperalgesia = 15 cm2 15 minutes after ID administration of 100 µg capsaicin.
* Demonstration of negative hyperalgesia as defined by an area of hyperalgesia < 5 cm2 15 minutes after ID administration of capsaicin vehicle.
* Subject with a skin type compatible with the measures, and without significant skin allergies, pigmentary disorders, or any active dermatological conditions that might interfere with the conduct of the study.

Exclusion Criteria:

* Subject has had a clinically significant illness in the 4 weeks before screening.
* Use of prescribed medications and herbal supplements in the 7 days prior to dosing or over the counter preparations, including multivitamins and paracetamol, in the 48 h before dosing.
* Subject has a significant history of drug/solvent abuse (within 2 years prior to Day 1), or a positive drugs of abuse test at screening.
* Subject with a history of alcohol abuse or currently drinks in excess of 28 units per week (males), or has a positive breath alcohol test at the Screening visit or on Day 1.
* Subject has a Heat pain tolerance threshold (HPTT) of = 50°C at screening.
* Subjects who do not develop erythema at the highest intensity of UV-B light used to establish Minimum erythema dose (MED).
* Known allergy or intolerance to capsaicin or hot peppers.
* Subjects who have any skin trauma, scars or other skin disorder or tattoos on their forearms or on the front of their thighs.
* Subject with active chronic pain conditions or a history of chronic pain conditions.
* Any condition that might interfere with the absorption, distribution, metabolism, and/or excretion of drugs.
* Previous ingestion of ICA-105665.
* Considering or scheduled to undergo any surgical procedure during the duration of the study.
* Prolonged QT/QTc interval (repeatedly = 450 msec). Received any agent known to alter hepatic or renal clearance (e.g., erythromycin, cimetidine, barbiturates, phenothiazines, clarithromycin, troleandomycin, ketoconazole, miconazole, fluconazole, itraconazole, etc.) for a period of 30 days prior to Day 1.
* History of risk factors for Torsades de Pointes (family history of long QT syndrome, heart failure, hypokalemia).
* Subject is unable to tolerate being blindfolded.
* Subject has participated in a clinical study involving capsaicin within 1 year of the Screening visit.
* Subject has a history of skin cancer.
* Subject has a clinically significant history of anemia.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2009-08; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Capsaicin: Visual Analogue Scale, hyperalgesia, allodynia, laser Doppler blood flow. UV-B pain assessments: Heat pain detection threshold, Heat pain tolerance threshold (HPTT), Laser Doppler blood flow (intensity and area), Skin temperature. | Capsaicin - Time 0, to 2 hours after injection. UV-B Pain: 2 hours post

SECONDARY OUTCOMES:
UV-B: Heat pain,Laser Doppler Blood Flow | 24 hours after irradiation

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- Pfizer Investigational Site, Wythenshawe, Manchester, United Kingdom
- Pfizer Investigational Site

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=ICA-105665-05&StudyName=Effects%20of%20ICA-105665%20Using%20the%20Intradermal%20Capsaicin%20and%20Ultraviolet%20B%20%28UV-B%29%20Models%20in%20Healthy%20Male%20Subjects